CLINICAL TRIAL: NCT03361397
Title: Effect of Nebulized Lidocaine on the Quality of Laryngeal Mask Airway Insertion: A Randomized, Double Blind, Controlled Study
Brief Title: Effect of Nebulized Lidocaine on the Quality of Laryngeal Mask Airway Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed galal aly, Assistant professor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17100246
Record Dates: First submitted 2017-11-24; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Airway Complication of Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine nebulization (Active Comparator): Inhalation of 10 mL nebulized lidocaine hydrochloride via mask nebulizer 5 min before laryngeal mask insertion.
  Interventions: Drug: Lidocaine Hydrochloride
- Distilled water nebulization (Placebo Comparator): Inhalation of 10 mL of nebulized distilled water solution via mask nebulizer 5 min before laryngeal mask insertion in the preoperative period.
  Interventions: Drug: Distilled Water

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — Lidocaine hydrochloride will be used via mask nebulizer before LMA insertion
  Other Names: Xylocaine
  Arms: Lidocaine nebulization
Drug: Distilled Water — Distilled Water will be used via mask nebulizer before LMA insertion
  Other Names: DW
  Arms: Distilled water nebulization

SUMMARY:
The primary outcome of this study will be the effect of lidocaine nebulization before LMA insertion on LMA insertion score (within 1 minute of LMA insertion) in adult patients undergoing surgery under general anesthesia.

The secondary outcome measures are the effect of LMA insertion on heart rate, arterial blood pressure, SpO2, the first time insertion rate of the LMA, and postoperative complications during LMA removal (soft tissue trauma, coughing, and laryngospasm).

DETAILED DESCRIPTION:
Patients will be randomly allocated into two groups of equal size to receive lidocaine nebulization, group L (GL) or distilled water nebulization, group W (GW/control). Randomization will be performed using GL and GW registers, which will be placed in sealed envelopes prior to study initiation and opened prior to anesthesia by a physician who will prepare the solution for nebulization and will identify it with the patient number, according to the envelope drawn. Group L patients (n = 40) will receive 10 mL lidocaine 4%, and GW patients (n = 40) will receive 10 mL distilled water (DW) by nebulizer mask 5 min prior to anesthesia. All patients will be preoxygenated with 100% oxygen for 3 minutes via mask gently placed over the face and thereafter Propofol 2.5 mg/kg slowly IV plus Fentanyl 1 µg/kg IV will be used for induction of anesthesia, and isoflurane for maintenance of anesthesia in both groups.

After confirming sufficient level of anesthesia (loss of eye lash reflex and jaw relaxation), the standard technique for LMA insertion (Brain,s method) will be used in both groups. Water based jelly will be applied on the posterior surface of the LMA and pressed along the palato-pharyngeal curve using the index finger. It is finally pushed further down till resistance is felt. A size 3 LMA will be used in women and a size 4 in men. Proper placement of LMA will be confirmed with bilateral equally audible breath sounds, chest movements and square wave capnography. Patients will be allowed to breathe spontaneously after successful LMA insertion.

The overall insertion condition will be assessed via a modified three point scale consisting of six variables, which include:

Mouth opening (3: full; 2: partial; 1: none) Ease of insertion (3: easy; 2: difficult; 1: impossible) Swallowing (3: nil; 2: slight; 1: gross) Coughing or gagging (3: nil; 2: slight; 1: gross) Head or limbs movement (3: nil; 2: slight; 1: gross), and Laryngospasm (3: nil; 2: partial; 1: total). Total score Insertion condition 18 Excellent 16-17 Satisfactory <16 Poor Any failure of insertion in both groups (defined as failure to insert the LMA after 3rd time), will be managed by endotracheal intubation.

At the end of the operation, LMA will be removed under deep anesthesia and replaced with Guedel's airway. Oxygen will be continued with a face mask until full recovery, and then the patients will be moved to the PACU.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (Age >18 yrs)
* ASA grade 1&2
* Scheduled to undergo various elective surgical procedures under general anesthesia using LMA.

Exclusion Criteria:

* Patients requiring endotracheal intubation
* Heavy smokers
* Grossly obese patients (Body mass index >35 kg/m2)
* Patients with suspected difficult airway (Mallampati Grade III or IV)
* Hypersensitivity to the used drugs
* Significant cardiovascular
* Significant pulmonary disease
* liver disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-11-30 (Estimated); Primary Completion 2018-04-02 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
LMA insertion score | within 1 minute of LMA insertion
  modified three point scale consisting of six variables, which measures the easiness of LMA insertion. Total score Insertion condition 18 Excellent 16-17 Satisfactory <16 Poor

SECONDARY OUTCOMES:
Heart rate | 1, 3, 5 minutes after LMA insertion
  Beat /min
Arterial blood pressure | 1, 3, 5 minutes after LMA insertion
  mm Hg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gupta A, Kaur S, Attri JP, Saini N. Comparative evaluation of ketamine - propofol, fentanyl - propofol and butorphanol-propofol on haemodynamics and laryngeal mask airway insertion conditions. J Anaesthesiol Clin Pharmacol. 2011 Jan;27(1):74-8. PMID 21804711
- [Background] Williams KA, Barker GL, Harwood RJ, Woodall NM. Combined nebulization and spray-as-you-go topical local anaesthesia of the airway. Br J Anaesth. 2005 Oct;95(4):549-53. doi: 10.1093/bja/aei202. Epub 2005 Aug 26. PMID 16126785